CLINICAL TRIAL: NCT00115388
Title: Community-Based Trial of Screening for Chlamydia Trachomatis to Prevent Pelvic Inflammatory Disease
Acronym: POPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Principal Investigator, Dr Pippa Oakeshott, Professor of General Practice, St George's, University of London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COHSR4PG
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Pelvic Inflammatory Disease; Chlamydia Infections
Keywords: Pelvic inflammatory disease; Chlamydia trachomatis; Screening
MeSH Terms: conditions — Pelvic Inflammatory Disease; Chlamydia Infections | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferred screening control group (Other): Samples from women in the control group were stored and tested at the end of the trial
  Interventions: Procedure: Screening for chlamydia using self-taken vaginal swabs

INTERVENTIONS:
Procedure: Screening for chlamydia using self-taken vaginal swabs — Women in the intervention group will be tested for chlamydia and those found to be infected will be referred for treatment and partner notification

SUMMARY:
Chlamydial infection is a common, sexually transmitted disease which women can have without knowing. Untreated, it can lead to an infection of the womb and fallopian tubes called pelvic inflammatory disease (PID), which can cause infertility. There has been only one trial of chlamydia screening and this was in American women in 1992 and used outdated tests. We now need to see if screening using modern tests and self-taken swabs works in a high risk, young, multiethnic female population in the United Kingdom (UK).

The study is a randomised trial. It will involve asking women students in college bars to complete confidential questionnaires on sexual health and to provide self-administered vaginal swabs. We have successfully done this in a small pilot study. Participants will be told that the tests are for research purposes only and that if they think they may have been at risk of a sexually transmitted infection they should get checked at a clinic. If the trial shows that chlamydia screening using these new methods prevents PID, extending this community-based intervention nationwide could improve women's reproductive health and wellbeing and might prevent some women from becoming infertile

DETAILED DESCRIPTION:
Background: Pelvic inflammatory disease (PID) is common and can lead to infertility, ectopic pregnancy or chronic pelvic pain.

Objectives: To see if screening and treatment of chlamydial infection reduces the incidence of PID over 12 months, and to investigate the natural history of chlamydial infection and the role of bacterial vaginosis (BV) in the development of chlamydia associated PID.

Design: Randomised trial over one year

Setting: Common rooms, bars and lecture theatres at universities and colleges in London, UK.

Participants: 2500 sexually active female students aged <28 years will be asked to complete a questionnaire on sexual health and to provide a self-administered vaginal swab and smear with follow up after a year.

Intervention: Following randomisation, vaginal swabs from intervention women will be tested for chlamydia by PCR and those infected referred for treatment. Vaginal swabs from control women will be stored and analysed after a year. Vaginal smears will be Gram stained and analysed for BV.

Main outcome measure: Incidence of clinical PID over 12 months in intervention and control groups.

Possible cases of PID will be identified from questionnaires and record searches. Confirmation of the diagnosis will be done by detailed review of medical records by two independent researchers blind to whether the woman is in the intervention or control group.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active

Exclusion Criteria:

* Never been sexually active
* Tested for chlamydia in past 3 months and no new sexual partner since then
* Pregnant

Ages: 16 Years to 27 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2531 (Actual)
Dates: Start 2004-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure in the complete cohort: Incidence of clinical PID over 12 months in intervention and control groups. | 12 months

SECONDARY OUTCOMES:
Secondary outcome measures after 12 months in women with chlamydial infection at baseline: | 12 months
Control group (untreated): | 12 months
Incidence of PID. | 12 months
Percentage with spontaneous clearance of genital infection. | 12 months
Relative risk of PID in women with and without BV | 12 months
3. Intervention group (treated): Reinfection rate. | 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Oakeshott, MD FRCP, Principal Investigator — St George's, University of London; Phillip Hay, FRCP, Study Chair — St George's, University of London
Locations (1):
- St George's Hospital Medical School, London, United Kingdom

REFERENCES:
- [Derived] Hay PE, Kerry SR, Normansell R, Horner PJ, Reid F, Kerry SM, Prime K, Williams E, Simms I, Aghaizu A, Jensen J, Oakeshott P. Which sexually active young female students are most at risk of pelvic inflammatory disease? A prospective study. Sex Transm Infect. 2016 Feb;92(1):63-6. doi: 10.1136/sextrans-2015-052063. Epub 2015 Jun 16. PMID 26082320
- [Derived] Oakeshott P, Kerry S, Aghaizu A, Atherton H, Hay S, Taylor-Robinson D, Simms I, Hay P. Randomised controlled trial of screening for Chlamydia trachomatis to prevent pelvic inflammatory disease: the POPI (prevention of pelvic infection) trial. BMJ. 2010 Apr 8;340:c1642. doi: 10.1136/bmj.c1642. PMID 20378636
- [Derived] Oakeshott P, Kerry S, Atherton H, Aghaizu A, Hay S, Taylor-Robinson D, Simms I, Hay P. Community-based trial of screening for Chlamydia trachomatis to prevent pelvic inflammatory disease: the POPI (prevention of pelvic infection) trial. Trials. 2008 Dec 10;9:73. doi: 10.1186/1745-6215-9-73. PMID 19077198
- [Derived] Atherton H, Banks D, Harbit R, Long L, Chadd F, Hay P, Kerry S, Simms I, Oakeshott P. Recruitment of young women to a trial of chlamydia screening - as easy as it sounds? Trials. 2007 Dec 4;8:41. doi: 10.1186/1745-6215-8-41. PMID 18053199